CLINICAL TRIAL: NCT06079281
Title: A Phase 3, Randomized, Double-blinded, Placebo-controlled, Multicenter Study to Evaluate Efficacy and Safety of ALXN1850 (Recombinant Alkaline Phosphatase) Administered Subcutaneously in Adolescent (12 to < 18 Years of Age) and Adult Participants With Hypophosphatasia Who Have Not Previously Been Treated With Asfotase Alfa
Brief Title: Phase 3 Study of ALXN1850 Versus Placebo in Adolescent and Adult Participants With HPP Who Have Not Previously Been Treated With Asfotase Alfa
Acronym: HICKORY
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Alexion Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D8590C00002; ALXN1850-HPP-301 (Other: Alexion Pharmaceuticals, Inc.)
Record Dates: First submitted 2023-10-06; First posted 2023-10-12 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Hypophosphatasia
Keywords: Hypophosphatasia; HPP; Asfotase Alfa; ALXN1850
MeSH Terms: conditions — Hypophosphatasia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Placebo Group (Placebo Comparator): During the Randomized Evaluation Period, the placebo group will receive placebo on Day 1, followed by once every 2 weeks (q2w) via SC injection for 24 weeks. Participants will enter the OLE Period and receive bodyweight dependent doses of either 20mg, 35mg, or 50mg of ALXN1850 and continue q2w dosing with ALXN1850 for up to 132 weeks.
  Interventions: Drug: Placebo
- ALXN1850 Group (Experimental): Starting at Day 1 of the Randomized Evaluation Period, the ALXN1850 group will receive bodyweight dependent doses of either 20mg, 35mg or 50mg of ALXN1850 once q2w via SC injection, for 24 weeks. Participants will enter the OLE Period and continue q2w dosing with ALXN1850 for up to 132 weeks.
  Interventions: Drug: ALXN1850; Drug: Placebo

INTERVENTIONS:
Drug: ALXN1850 — ALXN1850 will be administered via subcutaneous (SC) injection.
  Arms: ALXN1850 Group
Drug: Placebo — Placebo will be administered via SC injection.

SUMMARY:
The primary objective of this study is to assess the efficacy of ALXN1850 versus placebo on functional outcomes in adolescent and adult participants with HPP who have not previously been treated with asfotase alfa.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of HPP documented in the medical records
* Must meet 1 of the following criteria:

  1. Documented ALPL gene variant (pathogenic, likely pathogenic, or variant of unknown significance) from a Clinical Laboratory Improvement Amendments (CLIA) or ISO 15189 certified laboratory (Section 8.7 )
  2. Plasma PLP above the upper limit of normal (ULN) during the Screening Period (central or local laboratory results allowed per local regulations)
* Must meet 1 of the following criteria without a probably cause other than HPP:

  1. Serum ALP activity below the age- and sex-adjusted normal range during the screening period as measured by the Central Laboratory
  2. Two documented serum ALP activity results, at least 15 days apart, below the age- and sex-adjusted local laboratory normal range during the 24 months before the Day 1 Visit. Note: Local laboratories need to be CLIA or ISO 15189 certified, or have other local equivalent laboratory certification with Alexion's approval.
* Two separate 6MWTs at below 85% of the predicted distance (for age, sex, weight, and height) during the Screening Period without a probable cause other than HPP

Exclusion Criteria:

* History or presence of cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrinological, hematological, neurological disorders, or any other disorders that are capable of significantly altering the absorption, metabolism, or elimination of drugs; constituting a risk when taking the study intervention; or interfering with the interpretation of data as determined by the Investigator
* Diagnosis of primary or secondary hyperparathyroidism
* Hypoparathyroidism, unless secondary to HPP
* Any new fracture within 12 weeks before Day 1 (excluding pseudofractures)
* Planned surgical intervention which may impact the results of study assessments (in the opinion of the Investigator) during the Randomized Evaluation Period
* History of allergy or hypersensitivity to any ingredient contained in ALXN1850 or the placebo comparator (Table 9)

Ages: 12 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 124 (Actual)
Dates: Start 2024-01-03 (Actual); Primary Completion 2025-07-09 (Actual); Study Completion 2028-03-29 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in 6-Minute Walk Test (6MWT) at the end of the Randomized Evaluation Period (Day 169) | Baseline, Day 169

SECONDARY OUTCOMES:
Change from Baseline in 30-second Sit to Stand (STS) Test Score at the end of the Randomized Evaluation Period (Day 169) | Baseline, Day 169
Change from Baseline in Lower Extremity Functional Scale (LEFS) Score at the end of the Randomized Evaluation Period (Day 169) | Baseline, Day 169
Change from Baseline in BPI-SF pain severity score at the end of the Randomized Evaluation Period (Day 169) (adult cohort only) | Baseline, Day 169
Change from Baseline in FACIT-Fatigue score at the end of the Randomized Evaluation Period (Day 169) (adult cohort only) | Baseline, Day 169
Change from Baseline in Timed Up-and-Go (TUG) at the end of the Randomized Evaluation Period (Day 169) | Baseline, Day 169
Change from Baseline in Percent Predicted 6MWT at the end of the Randomized Evaluation Period (Day 169) | Baseline, Day 169
Radiographic Global Impression of Change (RGI-C) Score at the end of the Randomized Evaluation Period (Day 169) | Day 169
RGI-C Responder at the end of the Randomized Evaluation Period (Day 169) | Day 169
Change from Baseline in Rickets Severity Score (RSS) at the end of the Randomized Evaluation Period (Day 169) | Baseline, Day 169

CONTACTS AND LOCATIONS:
Locations (61):
- United States (5):
  - Research Site, Indianapolis, Indiana
  - Research Site, Garden City, New York
  - Research Site, Durham, North Carolina
  - Research Site, Columbus, Ohio
  - Research Site, Nashville, Tennessee
- Research Site, Ciudad de Buenos Aires, Argentina
- Australia (4):
  - Research Site, Clayton
  - Research Site, Herston
  - Research Site, Parkville
  - Research Site, St Leonards
- Brazil (5):
  - Research Site, Belo Horizonte
  - Research Site, Brasília
  - Research Site, Recife
  - Research Site, Salvador
  - Research Site, São Paulo
- Canada (5):
  - Research Site, Calgary, Alberta
  - Research Site, Edmonton, Alberta
  - Research Site, Winnepeg, Manitoba
  - Research Site, Oakville, Ontario
  - Research Site, Trois-Rivières, Quebec
- China (7):
  - Research Site, Beijing
  - Research Site, Changsha
  - Research Site, Chengdu
  - Research Site, Nanchang
  - Research Site, Qingdao
  - Research Site, Shanghai
  - Research Site, Shenzhen
- France (2):
  - Research Site, Paris
  - Research Site, Poitiers
- Germany (5):
  - Research Site, Bad Reichenhall
  - Research Site, Berlin
  - Research Site, Bonn
  - Research Site, Hamburg
  - Research Site, Würzburg
- Israel (2):
  - Research Site, Ashkelon
  - Research Site, Ramat Gan
- Italy (6):
  - Research Site, Florence
  - Research Site, Milan
  - Research Site, Padua
  - Research Site, Pisa
  - Research Site, San Giovanni Rotondo
  - Research Site, Verona
- Japan (5):
  - Research Site, Hiroshima
  - Research Site, Iizuka-shi
  - Research Site, Osaka
  - Research Site, Sapporo
  - Research Site, Yaizu-shi
- Research Site, Lodz, Poland
- South Korea (2):
  - Research Site, Seoul
  - Research Site, Suwon
- Spain (6):
  - Research Site, Barcelona
  - Research Site, Granada
  - Research Site, Madrid
  - Research Site, San Cristóbal de La Laguna
  - Research Site, Santander
  - Research Site, Vitoria-Gasteiz
- Taiwan (2):
  - Research Site, Taipei
  - Research Site, Taoyuan District
- Turkey (Türkiye) (2):
  - Research Site, Ankara
  - Research Site, Erzurum
- Research Site, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Alexion has a public commitment to allow requests for access to study data and will be supplying a protocol, CSR, and plain language summaries.
Supporting Information: Study Protocol, SAP, CSR

REFERENCES:
- See also: Routing the applicable forms for final approval prior to submission by the CTIS Expert — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D8590C00002&attachmentIdentifier=f48c8a4c-faf9-4dc8-bfaa-861cfae7f8ff&fileName=HPP-301_Structured_Data_Form_SM-1_(2).pdf&versionIdentifier=